CLINICAL TRIAL: NCT06969872
Title: The Effects of ABKefir on Functional Constipation in Subjects: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effects of Probiotics on Symptoms of Constipation in Adults With Functional Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: SYNBIO TECH INC. Kaohsiung Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS2-24134
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Functional Constipation (FC)
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): The composition of placebo capsules is same as the experimental capsules, except that they don't contain probiotics.
  Interventions: Dietary Supplement: Placebo
- Low dose of ABKefir (Experimental): Low dose of probiotics, 5×10^9 CFU/capsule
  Interventions: Dietary Supplement: Probiotics (ABKefir)
- High dose of ABKefir (Experimental): High dose of probiotics, 1×10^10 CFU/capsule
  Interventions: Dietary Supplement: Probiotics (ABKefir)

INTERVENTIONS:
Dietary Supplement: Placebo — Take a capsule of placebo within 30 minutes after breakfast, and once a day.
  Arms: Placebo
Dietary Supplement: Probiotics (ABKefir) — Take a capsule of ABKefir within 30 minutes after breakfast, and once a day.
  Arms: High dose of ABKefir; Low dose of ABKefir

SUMMARY:
The purpose of this study was to evaluate the efficacy of 1 capsules of ABKefir per day on symptoms of constipation in subjects with functional constipation by clinical trial.

DETAILED DESCRIPTION:
This randomized, placebo-controlled clinical trial will be conduct for 8 weeks with one hundred and sixty-five adults. Subjects will be recruited and randomly assigned into three groups: (1) placebo, n = 55; (2) low dose of ABKefir , n = 55; (3) high dose of ABKefir, n = 55. During the first 4 weeks of supplement, the subjects should take one capsule of placebo or ABKefir daily. Apart from containing no probiotics, the content of placebo is same as ABKefir. After that, the next 4 weeks is to have a follow-up of subjects. During this phase, subjects don't need to supplement. Subjects should complete the assessment of anthropometric measurement, defecation questionnaire , food record, feces and blood collection at week 0, 4 and week 8.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged 18-75 years old
* fulfill Rome IV criteria for functional constipation
* have not participated in similar research in the past three months

Exclusion Criteria:

* Personal or family history of colon cancer, celiac disease, and inflammatory bowel disease
* Irritable bowel syndrome diagnosed during colonoscopy
* Those who are pregnant recently (including men and women), or are pregnant or breastfeeding women.
* Taking antidepressants, anti-anxiety drugs and other psychotropic drugs.
* Long-term medication is required to improve constipation
* Those diagnosed with myocardial infarction, cerebral infarction, malignant tumor and/or other serious diseases are not suitable for participating in the study.
* Allergic symptoms to probiotics or any ingredients
* Having a history of serious mental illness
* Drug-related crimes or alcohol problems
* Have recently traveled to areas where parasitic diseases are prevalent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline symptoms of constipation at week 4 and 8 | Week 0, 4 and 8
  Compared the difference of bowel movements between the week 0, 4 and 8.
Change from baseline symptoms of constipation at week 4 and 8 | Week 0, 4 and 8
  Compared the difference of stool consistency between the week 0, 4 and 8.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Chi Pan, MS student, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, South, Taiwan